CLINICAL TRIAL: NCT00001667
Title: Genotype/Phenotype Correlation of Movement Disorders and Other Neurological Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970097; 97-N-0097
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-02

CONDITIONS: Movement Disorders; Myoclonus; Nervous System Diseases; Tic Disorders; Tremor
Keywords: Family Studies; Genetic; Myoclonus; Tics; Tremor; Movement Disorders; Neurological Disease
MeSH Terms: conditions — Movement Disorders; Myoclonus; Nervous System Diseases; Tic Disorders; Tremor; Tics

SUMMARY:
The purpose of this protocol is to identify families with inherited neurologic conditions, especially movement disorders, to evaluate affected and unaffected individuals clinically, and to obtain blood samples for genetic analysis.

DETAILED DESCRIPTION:
The purpose of this protocol is to identify families with inherited neurologic conditions, especially movement disorders, to evaluate affected and unaffected individuals clinically, and to obtain blood samples for genetic analysis.

ELIGIBILITY:
Neurologic disease or movement disorders affecting 2 or more family members.

No conditions in which phlebotomy is contra-indicated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 1997-03; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Higgins JJ, Nee LE, Vasconcelos O, Ide SE, Lavedan C, Goldfarb LG, Polymeropoulos MH. Mutations in American families with spinocerebellar ataxia (SCA) type 3: SCA3 is allelic to Machado-Joseph disease. Neurology. 1996 Jan;46(1):208-13. doi: 10.1212/wnl.46.1.208. PMID 8559377
- [Background] Silveira I, Lopes-Cendes I, Kish S, Maciel P, Gaspar C, Coutinho P, Botez MI, Teive H, Arruda W, Steiner CE, Pinto-Junior W, Maciel JA, Jerin S, Sack G, Andermann E, Sudarsky L, Rosenberg R, MacLeod P, Chitayat D, Babul R, Sequeiros J, Rouleau GA. Frequency of spinocerebellar ataxia type 1, dentatorubropallidoluysian atrophy, and Machado-Joseph disease mutations in a large group of spinocerebellar ataxia patients. Neurology. 1996 Jan;46(1):214-8. doi: 10.1212/wnl.46.1.214. PMID 8559378
- [Background] Ichinose H, Ohye T, Matsuda Y, Hori T, Blau N, Burlina A, Rouse B, Matalon R, Fujita K, Nagatsu T. Characterization of mouse and human GTP cyclohydrolase I genes. Mutations in patients with GTP cyclohydrolase I deficiency. J Biol Chem. 1995 Apr 28;270(17):10062-71. doi: 10.1074/jbc.270.17.10062. PMID 7730309